CLINICAL TRIAL: NCT06997536
Title: Comparison of Postoperative Analgesic Efficacy of Ultrasound-Guided Ilioinguinal-Iliohypogastric Block, Transversus Abdominis Plane Block, and Quadratus Lumborum Block in Inguinal Hernia Surgery: A Prospective, Randomized Controlled Trial
Brief Title: Comparison of Postoperative Analgesic Efficacy of Ultrasound-Guided Ilioinguinal-Iliohypogastric Block, Transversus Abdominis Plane Block, and Quadratus Lumborum Block in Inguinal Hernia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ahmet Gültekin, Associate Professor, Namik Kemal University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: NamikKU-AGultekin-Meltem2025
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Inguinal Hernia; Transversus Abdominis Plane (TAP) Block; Iliohypogastric/Ilioinguinal Nerve Block; Quadratus Lumborum Block
Keywords: Inguinal hernia; Ilioinguinal-iliohypogastric block; Transversus abdominis plane block; Quadratus lumborum block
MeSH Terms: conditions — Hernia, Inguinal; Bites and Stings | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ilioinguinal/Iliohypogastric Block (Experimental): After spinal anesthesia was applied, a preoperative ilioinguinal/iliohypogastric block was administered to the side to be operated on.
  Interventions: Procedure: Ilioinguinal/iliohypogastric Nerve Block
- Transversus abdominis plane (TAP) block (Experimental): After spinal anesthesia was applied, a preoperative transversus abdominis plane (TAP) block was administered to the side to be operated on.
  Interventions: Procedure: Transversus abdominis plane (TAP) block
- Quadratus Lumborum Block (Experimental): After spinal anesthesia was applied, a preoperative quadratus lumborum block (QLB) was administered to the side to be operated on.
  Interventions: Procedure: Quadratus Lumborum Block (QLB)
- Control (No Intervention): No block was applied after spinal anesthesia.

INTERVENTIONS:
Procedure: Ilioinguinal/iliohypogastric Nerve Block — The aim of this study is to compare the analgesic efficacy of IL/IH block, TAP block, and QLB applied in inguinal hernia cases operated under spinal anesthesia, with each other and with a control group that did not receive any additional block to spinal anesthesia.
  Arms: Ilioinguinal/Iliohypogastric Block
Procedure: Transversus abdominis plane (TAP) block — The aim of this study is to compare the analgesic efficacy of IL/IH block, TAP block, and QLB applied in inguinal hernia cases operated under spinal anesthesia, with each other and with a control group that did not receive any additional block to spinal anesthesia.
  Arms: Transversus abdominis plane (TAP) block
Procedure: Quadratus Lumborum Block (QLB) — The aim of this study is to compare the analgesic efficacy of IL/IH block, TAP block, and QLB applied in inguinal hernia cases operated under spinal anesthesia, with each other and with a control group that did not receive any additional block to spinal anesthesia.
  Arms: Quadratus Lumborum Block

SUMMARY:
Inguinal hernia is a common condition, particularly among male patients, and represents one of the most frequent indications for lower abdominal surgeries. Postoperative acute pain and, more importantly, the progression of acute pain into chronic pain, remain significant challenges in the postoperative period. Effective postoperative pain management is therefore crucial in inguinal hernia repair.

In addition to systemic analgesia, various regional anesthesia techniques are employed in this setting. In recent years, peripheral nerve blocks such as the ilioinguinal-iliohypogastric (IL/IH) block, transversus abdominis plane (TAP) block, and quadratus lumborum block (QLB) have gained popularity for postoperative analgesia. These techniques offer several advantages, including reduced opioid consumption and decreased need for additional analgesics, while also minimizing hemodynamic instability and facilitating early mobilization.

The IL/IH block is performed by injecting a local anesthetic into the fascial plane between the transversus abdominis and internal oblique muscles, targeting the ilioinguinal and iliohypogastric nerves, which are branches of the L1 spinal nerve. The TAP block, first described by Rafi in 2001, involves injecting local anesthetic into the fascial plane between the internal oblique and transversus abdominis muscles within the Petit triangle, where the T6-T11 spinal nerve branches responsible for abdominal wall innervation are located. The quadratus lumborum block (QLB) was initially described by Blanco. The first version, known as QLB1, involves posterior injection of local anesthetic lateral to the quadratus lumborum muscle. In 2013, Jens Børglum introduced the transmuscular variant (QLB3), where the local anesthetic is administered between the quadratus lumborum and psoas muscles.

In this study, we aimed to compare postoperative outcomes in patients undergoing inguinal hernia repair under spinal anesthesia, with and without additional peripheral nerve blocks (IL/IH block, TAP block, and QLB). Specifically, we evaluated pain levels using the Visual Analog Scale (VAS) at the 30th minute, 2nd, 6th, 12th, and 24th hours postoperatively. We also assessed opioid-related side effects such as nausea and vomiting associated with patient-controlled analgesia (PCA) using tramadol, the total bolus and infusion doses of tramadol administered, and the amount of additional analgesia in the form of paracetamol. These outcomes were compared among the different block groups and with a control group that received only spinal anesthesia without any additional block.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as ASA I and II
* Patients aged 18 to 75 years
* Patients undergoing unilateral inguinal hernia surgery under spinal anesthesia

Exclusion Criteria:

* Patients with preoperative neurological sequelae
* Patients with a BMI >30
* Patients who refused to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score | Postoperative 30th minute, 2nd, 6th, 12th and 24th hours
  Postoperative pain will be assessed using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (the worst imaginable pain). Pain scores will be recorded at predefined time points during rest and movement.

SECONDARY OUTCOMES:
Total Opioid Consumption at 24 Hours. | At the end of the 24th hour
  For patient-controlled analgesia, tramadol 300 mg was prepared in 100 cc of isotonic saline with a concentration of 3 mg/cc. The infusion rate was set at 3 mL/hour, with a 5 mL bolus dose, a lock-out time of 4 hours, and the device was set to be used for 24 hours. In patients with a VAS score of 4 or higher despite opioid demand from the patient-controlled analgesia device, an additional 1 gram of IV paracetamol was planned to be administered as an adjunct analgesic. Total infusion and bolus doses of tramadol over 24 hours were recorded.

OTHER OUTCOMES:
Total nausea and vomiting count over 24 hours | At the end of the 24th hour
  The number of nausea and vomiting episodes experienced by the patients over 24 hours was recorded.
Need for additional analgesia | At the end of the 24th hour
  In patients with a VAS score of 4 or higher despite opioid requests via the patient-controlled analgesia device, 1 gram of IV paracetamol was planned to be administered as an additional analgesic. At the end of the 24th postoperative hour, the total need for additional analgesia was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Namik Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No